CLINICAL TRIAL: NCT02185963
Title: Effect of Rosuvastatin on Function of High Density Lipoprotein Cholesterol in Patients With Type 2 Diabetes
Brief Title: Effect of Rosuvastatin on Function of High Density Lipoprotein Cholesterol in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNUBH_ENDO05
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes
Keywords: Diabetes; Dyslipidemia; HDL function; Cholesterol efflux; MCA assay; MCP-1
MeSH Terms: conditions — Diabetes Mellitus; Dyslipidemias | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rosuvastatin (Experimental): Rosuvastatin will be started in type 2 DM and having 1 or more cardiovascular risk factors
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20mg once a daily for 12 weeks
  Other Names: Crestor

SUMMARY:
The patients who have achieved LDL-C levels below the currently recommended targets may still experience cardiovascular events. To reduce further the risk of coronary heart disease (CHD), raising HDL-C and lowering TG may be the secondary therapeutic target. However, increased HDL-C levels do not mean increase in functional HDL-C. It also remains controversial whether functional HDL is more important than total circulating levels of HDL-C in reducing CHD.

Actually, the increased concentration of HDL alone might be ineffective indicating that qualitative changes in HDL levels in response to drug interventions are required to result in clinical benefit.

The investigators set up a clinical trial investigating effect of (rosuva)statin treatment on functional HDL-C levels particularly in Asian populations, who have relatively low HDL-C.

DETAILED DESCRIPTION:
1. Study design Study subject Number of Subjects (N = 30)
2. Study outcome

   Primary outcome - functional HDL-C Secondary outcome - Non-HDL cholesterol
3. Evaluation of functional aspect of HDL Cholesterol efflux from macrophages LDL-induced monocyte chemotactic activity (MCA) Assay Quantitation of gene expression of monocyte chemotactic protein-1 (MCP-1)

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes
2. HbA1c ≥ 7.5%
3. Age ≥ 30
4. low HDL-C (<40 mg/dl in men or <50 mg/dl in women) and having 1 or more risk factors: 1) Body mass index (BMI) ≥ 25 kg/m2 (overweight); 2) LDL-C level ≥ 130 mg/dl; 3) TG level ≥150 mg/dl; 4) Systolic blood pressure (SBP)/diastolic blood pressure (DBP) ≥140/90 mmHg or taking antihypertensive medication; 5) Current smoker; 6) Family history of CHD.

Exclusion Criteria:

1. Contraindication to rosuvastatin
2. Pregnant or breast feeding women
3. Reproductive-age women who refuse contraception
4. Type 1 diabetes, gestational diabetes, or diabetes with secondary cause
5. Chronic hepatitis B or C (except healthy carrier of HBV), liver disease (AST/ALT > 3-fold the upper limit of normal)
6. Renal failure (Cr > 2.0)
7. Cancer within 5 years (except squamous cell cancer, cervical cancer, thyroid cancer with appropriate treatment)
8. Not appropriate for lipid lowering treatment
9. Medications which affect glycemic control
10. Diseases which affect efficacy and safety of statin
11. Other clinical trial within 30 days

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Functional HDL-C | 12 weeks
  1. Cholesterol efflux from macrophages
  2. LDL-induced monocyte chemotactic activity (MCA) Assay
  3. Quantitation of gene expression of monocyte chemotactic protein-1 (MCP-1)

SECONDARY OUTCOMES:
Non-HDL-cholesterol = total cholesterol - HDL-C | 12 weeks
Patients with LDL-C < 70 mg/dl and HDL > 40 mg/dl in men; > 50 in women | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, PHD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Kim KM, Jung KY, Yun HM, Lee SY, Oh TJ, Jang HC, Lim S. Effect of rosuvastatin on fasting and postprandial endothelial biomarker levels and microvascular reactivity in patients with type 2 diabetes and dyslipidemia: a preliminary report. Cardiovasc Diabetol. 2017 Nov 9;16(1):146. doi: 10.1186/s12933-017-0629-0. PMID 29121934 (Retraction: PMID 30876421 Cardiovasc Diabetol. 2019 Mar 16;18(1):32)